CLINICAL TRIAL: NCT05939596
Title: Randomized, Blinded, Placebo-controlled Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of SARS-CoV-2 Bivalent mRNA Vaccine (LVRNA021) in Participants Aged 18 Years and Older Who Have Received SARS-CoV-2 Vaccine
Brief Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of SARS-CoV-2 Bivalent mRNA Vaccine (LVRNA021)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AIM Vaccine Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LVRNA021-I-01
Record Dates: First submitted 2023-07-07; First posted 2023-07-11 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SARS-CoV-2 Bivalent mRNA Vaccine (LVRNA021) (Experimental): 100 μg /1.0 mL/dose, One booster dose 1.0mL IM injection of SARS-CoV-2 Bivalent mRNA Vaccine (LVRNA021).
  Interventions: Biological: SARS-CoV-2 Bivalent mRNA Vaccine
- Saline (Placebo Comparator): One booster dose 1.0mL IM injection of saline.
  Interventions: Other: Saline

INTERVENTIONS:
Biological: SARS-CoV-2 Bivalent mRNA Vaccine — 100 μg /1.0 mL/dose, slightly milky white and clear liquid, intramuscular injection into the lateral deltoid muscle of the upper arm.
  Other Names: LVRNA021
  Arms: SARS-CoV-2 Bivalent mRNA Vaccine (LVRNA021)
Other: Saline — 100 μg /1.0 mL/dose, intramuscular injection into the lateral deltoid muscle of the upper arm.
  Arms: Saline

SUMMARY:
This trial is a phase I clinical trial of a SARS-CoV-2 Bivalent mRNA Vaccine (LVRNA021). The trial used a randomized, blinded, placebo-controlled design to evaluate the safety, tolerability, and preliminary immunogenicity of the trial vaccine in participants Aged 18 Years and Older who had received SARS-CoV-2 Vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 years and older, both male and female, who can provide legal identity certificate of participants;
2. The subject understands the contents of the Informed Consent Form and the vaccination situation of this vaccination, voluntarily signs the Informed Consent Form, and has the ability to use the thermometer, scale and fill in the Diary Card and Contact Card as required (if the subject is unable to sign the Informed Consent Form by himself/herself due to limited reading and writing ability, the informed consent form and signature of the Informed Consent Form can be completed under the witness' s witness);
3. Able to communicate well with investigators and understand and comply with the requirements of this trial;
4. Completion of basic immunization with SARS-CoV-2 vaccine ≥ 6 months;
5. Negative nucleic acid test for SARS-CoV-2 within 3 days prior to vaccination;
6. Women who have used effective contraception within 2 weeks prior to inclusion in this trial, have a negative pregnancy test (pregnancy test can be exempted for those who have been amenorrheic for at least 1 year or have a documented history of surgical sterilization), and voluntarily agree to continue using at least 1 effective contraception within 6 months after vaccination [effective contraception includes: oral contraceptives, injected or implanted contraception, sustained-release local contraceptives, hormonal patches, intrauterine device (IUD), sterilization, abstinence, condoms (men), diaphragms, cervical caps, etc.];
7. Healthy participants or participants with mild underlying disease [stable condition without worsening (requiring no hospitalization or major modification of treatment regimen, etc.) for at least 3 months prior to inclusion in this trial].

Exclusion Criteria:

1. Abnormal blood routine, blood biochemistry, coagulation routine, D-dimer, troponin, urine routine and other clinical test indicators during the screening period, and the investigator judges that the health condition is uncertain and further diagnosis is required, or the investigator judges that the patient is not suitable for vaccination in combination with the medical history and clinical manifestations;
2. Body mass index (BMI) <18 kg/m 2 or >30 kg/m 2;
3. Individuals with any infectious disease, acute infection, acute phase of chronic infection (such as active untreated pulmonary tuberculosis, etc.) or any advanced immune disease (inquiry);
4. Infected within last 6 months or likely infected with SARS-CoV-2;
5. Positive HIV test result at screening;
6. Fever on the day of investigational vaccination (axillary temperature ≥ 37.3℃) or within 3 days, or use of antipyretic and analgesic drugs within 3 days;
7. Women with a positive pregnancy test (surgical sterilizers who are menstruating or amenorrheic for at least 1 year or have medical records may be exempted from pregnancy testing), or breastfeeding women, or women planning to become pregnant from screening through 6 months after booster vaccination, men whose partners plan to become pregnant, or plan to donate sperm and eggs;
8. Previous history of allergic or allergic reactions to vaccines or drugs, such as urticaria, severe skin eczema, dyspnea, laryngeal edema, angioneurotic edema, etc.;
9. Administration of any vaccine within 28 days prior to booster vaccination with investigational vaccine;
10. Have participated within 28 days prior to booster vaccination with investigational vaccine or plan to participate in other drug clinical trials within 12 months after booster vaccination;
11. Patients with a history of thrombocytopenia or other coagulation disorders, which may cause contraindications to subcutaneous blood sampling or injection, and patients with a history of thrombosis;
12. Known history or diagnosis of diseases affecting immune system function, such as cancer (except basal cell carcinoma of the skin), congenital or acquired immunodeficiency, uncontrolled autoimmune diseases, etc. (such as systemic lupus erythematosus, autoimmune thyroid disease, multiple sclerosis);
13. Absence of spleen or functional absence of spleen;
14. Chronic use (≥14 consecutive days) of immunosuppressants or other immunomodulatory drugs (eg, corticosteroids: prednisone or drugs of the same class) within 6 months prior to booster vaccination with the investigational vaccine, but topical medications (eg, ointments, eye drops, inhalers, or nasal sprays) are allowed and should not exceed the dose recommended in the package insert;
15. Immunoglobulins and/or blood products received within 3 months prior to the investigational booster vaccination;
16. Suspected or known alcohol dependence or drug abuse that could compromise the safety evaluation or subject compliance;
17. Other conditions that the investigator considers inappropriate for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of solicited and unsolicited adverse events | 0-28 days after booster vaccination.
  Incidence of solicited and unsolicited adverse events 0-28 days after booster vaccination in all participants.

SECONDARY OUTCOMES:
Incidence of abnormal laboratory-related parameters | 3 days after booster vaccination
  Incidence of abnormal laboratory-related parameters on the third day after booster vaccination in participants.
Incidence of serious adverse events (SAEs) and adverse events of special interest (AESIs) | Within 12 months after booster vaccination.
  Incidence of serious adverse events (SAEs) and adverse events of special interest (AESIs) within 12 months after booster vaccination in all participants.
GMT, SCR, and GMI of neutralizing antibodies against SARS-CoV-2 (Delta, Omicron BA.5, XBB, and current major circulating strains) | 7, 14, 28 days after booster vaccination.
  GMT, SCR, and GMI of neutralizing antibodies against SARS-CoV-2 (Delta, Omicron BA.5, XBB, and current major circulating strains) on days 7, 14, and 28 after booster vaccination in participants.
GMT of neutralizing antibodies against SARS-CoV-2 (Delta, Omicron BA.5, XBB, and current major circulating strains) | 3, 6, 12 months after booster vaccination.
  GMT of neutralizing antibodies against SARS-CoV-2 (Delta, Omicron BA.5, XBB, and current major circulating strains) at months 3, 6, and 12 after booster vaccination in participants.
GMC, SCR, and GMI of IgG antibodies against S proteins of SARS-CoV-2 (Delta, Omicron BA.5, XBB, and current major circulating strains) | 7, 14, 28 days after booster vaccination.
  GMC, SCR, and GMI of IgG antibodies against S proteins of SARS-CoV-2 (Delta, Omicron BA.5, XBB, and current major circulating strains) on days 7, 14, and 28 after booster vaccination.
GMC of IgG antibodies against S proteins of SARS-CoV-2 (Delta, Omicron BA.5, XBB, and current major circulating strains) | 3, 6, 12 months after booster vaccination.
  GMC of IgG antibodies against S proteins of SARS-CoV-2 (Delta, Omicron BA.5, XBB, and current major circulating strains) at 3, 6, and 12 months after booster vaccination.

OTHER OUTCOMES:
Specific T cell responses secreting IL-2, IL-4, IL-13, IFN-γ cytokines (ELISpot assay) | 7, 14, 28 days after booster vaccination.
  Specific T cell responses secreting IL-2, IL-4, IL-13, IFN-γ cytokines (ELISpot assay) on days 7, 14, and 28 after booster vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: fan zhang, Study Director — AIM Vaccine Co., Ltd.
Locations (1):
- First Affiliated Hospital Bengbu, Bengbu, Anhui, China